CLINICAL TRIAL: NCT06662435
Title: A Pilot and Mixed-Methods Study of GYNecologic Cancer-Related COGnitive Impairment
Brief Title: GYNecologic Cancer-Related COGnitive Impairment
Acronym: GYNCOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Friends of Prentice (Other)
Responsible Party: Principal Investigator, Emma Barber, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00222610
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Cervical Cancers; Vulvar Cancers; Uterine Cancer; Cervix Cancer; Ovary Cancer
Keywords: cognitive impairment; gynecologic cancer; cancer related cognitive impairment
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Uterine Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GYNCOG Intervention (Experimental): Participants in the GYNCOG arm will be asked to participate in a home-based cognitive training program utilizing BrainHQ on study-provided tablets.
  Interventions: Behavioral: GYNCOG
- Control Group (No Intervention): Patients in the Control Group arm will receive usual care with no cognitive intervention.

INTERVENTIONS:
Behavioral: GYNCOG — Participants in the GYNCOG arm will be asked to participate in a home-based cognitive training program utilizing BrainHQ. Participants will be instructed to use the Brain HQ app for approximately 2.5 hours per week. Patients will be provided with a calendar to help keep track of daily BrainHQ use, including the number of exercises completed and the amount of time spent on the app per day.
  Patients will be asked to undergo the exercises that target the speed and accuracy of information processing. Examples of the exercises include:
  Double Decision: This exercise tests your ability to quickly identify and choose between two options.
  Eye for Detail: It challenges participants to spot small differences between two similar images.
  Participants will be asked to train approximately 30 minutes per BrainHQ session, 5 times per week (i.e., 2.5 hours per week) for 10 weeks, for a total of approximately 25 hours.
  Arms: GYNCOG Intervention

SUMMARY:
The goal of this study is to test a home-based and patient-tailored cognitive training intervention among gynecologic cancer patients who have completed chemotherapy and who have experienced cancer-related cognitive impairment.

DETAILED DESCRIPTION:
Gynecologic cancers are prevalent and long-term survivorship is increasing. In the United States, survivors of gynecologic cancer number over one million individuals and constitute more than 10% of all cancer survivors. Curative treatment usually involves systemic chemotherapy.

A distressing long-term side effect of cytotoxic chemotherapy is cancer-related cognitive impairment (CRCI), or "chemo brain," which has been reported to be present in up to 75% of patients and can linger for months or even decades after chemotherapy treatment. Despite increasing prevalence, patients report that CRCI has not been a focus of assessment or treatment, and the lack of understanding from providers has led to patient disempowerment. Within gynecologic oncology, CRCI is under-reported and understudied with no established effective treatment.

There is no currently established standard of care for managing CRCI in cancer survivors. However, existing literature highlights cognitive training as a promising nonpharmacological intervention. Cognitive training programs consist of structured cognitive exercises designed to target specific cognitive domains. It is postulated to engage neuroplasticity mechanisms, promote the formation of new neural connections, enhance cognitive reserve, and subsequently improve cognitive function and mitigate impairment. Clinically, cognitive training interventions have been shown to not only ameliorate subjective concerns but also improve objective cognitive function, such as memory and attention. It has also been associated with improved daily functioning and physical function.

The BrainHQ (Posit Science®) is an adaptive cognitive training program that addresses CRCI through scientifically validated exercises and an adaptive algorithm targeting memory, attention, and processing speed. The program's efficacy has been documented in diverse settings, including breast cancer survivors. Despite its use in other populations, cognitive training's potential in gynecologic oncology patients is unexplored.

This study will enroll patients with advanced gynecologic cancers who have completed adjuvant chemotherapy and are currently in surveillance with at least stable disease. Patients will be included if they screen positive for subjective report of cognitive impairment. This project will provide important, currently unknown information on the feasibility and acceptability of a cognitive training intervention in patients with advanced gynecologic cancers who report cognitive impairment following primary systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female; ≥18 years of age
* Presents to clinic with a confirmed diagnosis of a gynecologic cancer (e.g., ovarian, endometrial, cervical, or vulvar cancer) who have completed adjuvant chemotherapy with at least stable disease at time of screening.
* Screen positive for subjective cognitive impairment by answering affirmatively to at least one of three screener questions
* Fluent in spoken and written English
* Have access to the internet to complete assessments

Exclusion Criteria:

* Patients who have not received chemotherapy
* Patients with pre-existing neuropsychiatric disorders that would impact cognitive function, such as dementia, Alzheimer's disease, and schizophrenia.
* Patients with non-gynecologic causes of incurable metastatic cancers.
* Patients undergoing active interventions in other cognitive trials or patients currently using cognitive training programs such as Brain HQ, Luminosity, Elevate, Peak, Fit Brains, or CogniFit.
* Patients with self-report of learning disability or an unwillingness to participate in technology-based cognitive training programs.
* Pregnant women or prisoners
* Patients with impaired-decision making capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assessment Compliance | 20 weeks
  Assessment compliance will be defined as completing the cognitive assessments at baseline and at 10 weeks. The study will be considered feasible in terms of assessment compliance if at least 65% of all patients are compliant.
Adherence | 10 weeks
  Adherence will be defined as completing ≥80% of intended BrainHQ exercises over 10 weeks. The intervention would be considered not feasible if ≤ 28/40 of patients are considered adherent.

SECONDARY OUTCOMES:
Acceptability | 10 weeks
  Acceptability will be measured at the end of the intervention period using the Acceptability of Intervention Measure, a validated 4-item measure of perceived intervention acceptability. Total score ranges from 4-20, with higher scores indicating greater acceptability.
Change in Patient Reported Cognitive Function | 20 weeks
  Cognitive function will be measured via the Patient-Reported Outcomes Measurement Information System short-form on cognitive function. Each item on the measure is rated on a 5-point scale with a range in score from 6 to 30 with higher scores indicating greater cognitive impairment.
Change in Objective Cognitive Function | 20 weeks
  Objective cognitive function will be measured via the Montreal Cognitive Assessment-Blind version 8. This is a modified version of the standard Montreal Cognitive Assessment, which is designed to be used in situations where visual components of cognitive testing are not feasible and useful for testing in remote settings. The MoCA is a widely used screening tool for detecting cognitive impairment, assessing domains like memory, attention, language, and executive function. Total score ranges from 0-22, with higher scores indicating greater cognitive function.
Change in Physical Function | 20 weeks
  Physical function will be measured via the Patient-Reported Outcomes Measurement Information System short-form on physical function. Each item on the measure is rated on a 5-point scale with a range in score from 4 to 20 with lower scores indicating greater physical function.
Change in Fatigue | 20 weeks
  Fatigue will be measured via the Patient-Reported Outcomes Measurement Information System short-form on fatigue. Each item on the measure is rated on a 5-point scale with a range in score from 4 to 20 with higher scores indicating greater fatigue.
Change in Illness Impact on Social Roles and Daily Tasks | 20 weeks
  This will be measured via the Patient-Reported Outcomes Measurement Information System short-form on illness impact on social roles and daily tasks. Each item on the measure is rated on a 5-point scale with a range in score from 4 to 20 with higher scores indicating greater satisfaction in performing daily tasks.
Change in Sleep Disturbance | 20 weeks
  Sleep disturbance will be measured via the Patient-Reported Outcomes Measurement Information System short-form on sleep disturbance. Each item on the measure is rated on a 5-point scale with a range in score from 4 to 20 with higher scores indicating greater sleep disturbance.
Change in Depression | 20 weeks
  Depression will be measured via the Patient-Reported Outcomes Measurement Information System short-form on depression. Each item on the measure is rated on a 5-point scale with a range in score from 4 to 20 with higher scores indicating greater depression.
Change in Anxiety | 20 weeks
  Anxiety will be measured via the Patient-Reported Outcomes Measurement Information System short-form on anxiety. Each item on the measure is rated on a 5-point scale with a range in score from 4 to 20 with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barber, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No